CLINICAL TRIAL: NCT05230511
Title: Intravesical Lactobacillus rhamnosusGG Versus Saline Bladder Wash: A Randomized, Controlled, Comparative Effectiveness Clinical Trial
Brief Title: Intravesical LGG VS Saline Bladder Wash RCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00004287
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injuries; Neurogenic Bladder
Keywords: Intermittent Catheter
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic

STUDY DESIGN:
Intervention Model Description: Randomized, controlled comparative effectiveness clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Intravesical Lactobacillus RhamnosusGG and Bladder Wash (Treatment Phase) (Experimental): LGG® (Culturelle Probiotic LGG®) will be used. This is the product we have used in the past and for which we have demonstrated safety, tolerability, and preliminary efficacy. For the LGG® instillation in response to trigger symptoms, participants will be instructed to mix the contents of 1 LGG® capsule into 45 cc sterile 0.9% saline. After mixing, participants will draw up the 45cc liquid LGG® mixture into a 60cc syringe and instill via the intermittent catheter after the last catheterization prior to going to bed. Participants will be asked to return any remaining capsules at the end of the study. Participants will be instructed to complete the USQNB-IC at the time of symptoms (in real time) and daily during instillations for 2 days after the final instillation. Subjects will remain in this phase 6 months.
  Interventions: Drug: Lactobacillus RhamnosusGG
- Intravesical Bladder Wash (Treatment Phase) (Other): Participants will draw up the 45cc of normal saline into a 60cc syringe and instill via the intermittent catheter after the last catheterization prior to going to bed after trigger symptoms occur. Participants will be instructed to complete the USQNB-IC at the time of symptoms (in real time) and daily during instillations for 2 days after the final instillation. Subjects will remain in this phase 6 months.
  Interventions: Drug: Saline bladder wash
- Intravesical Lactobacillus RhamnosusGG and Bladder Wash (Prophylaxis Phase) (Experimental): LGG® (Culturelle Probiotic LGG®) will be used. This is the product we have used in the past and for which we have demonstrated safety, tolerability, and preliminary efficacy. For the LGG® instillation in response to trigger symptoms, participants will be instructed to mix the contents of 1 LGG® capsule into 45 cc sterile 0.9% saline. After mixing, participants will draw up the 45cc liquid LGG® mixture into a 60cc syringe and instill via the intermittent catheter after the last catheterization prior to going to bed. They will then instill the LGG® mixture every 2 days for the remainder of the 6 months. Participants will be asked to return any remaining capsules at the end of the study. Participants will be instructed to complete the USQNB-IC at the time of symptoms (in real time) and biweekly post-instillation. Subjects will remain in this phase 6 months.
  Interventions: Drug: Lactobacillus RhamnosusGG
- Intravesical Bladder Wash (Prophylaxis Phase) (Other): Participants will draw up the 45cc of normal saline into a 60cc syringe and instill via the intermittent catheter after the last catheterization prior to going to bed after trigger symptoms occur. They will then instill the saline BW every 2 days for the remainder of the 6 months. Participants will be instructed to complete the USQNB-IC at the time of symptoms (in real time) and biweekly post-instillation. Subjects will remain in this phase 6 months.
  Interventions: Drug: Saline bladder wash

INTERVENTIONS:
Drug: Lactobacillus RhamnosusGG — LGG® (Culturelle Probiotic LGG®) will be used. This is the product we have used in the past and for which we have demonstrated safety, tolerability, and preliminary efficacy. For the LGG® instillation, participants will be instructed to mix the contents of 1 LGG® capsule into 45 cc sterile 0.9% saline. After mixing, participants will draw up the 45cc liquid LGG® mixture into a 60cc syringe and instill via the intermittent catheter after the last catheterization prior to going to bed. Participants will be asked to return any remaining capsules at the end of the study. Participants will be instructed to complete the USQNB-IC at the time of symptoms (in real time), and then continue completing the USQNB-IC at the determined frequency for the phase.
  Other Names: Culturelle Probiotic LGG®
  Arms: Intravesical Lactobacillus RhamnosusGG and Bladder Wash (Prophylaxis Phase); Intravesical Lactobacillus RhamnosusGG and Bladder Wash (Treatment Phase)
Drug: Saline bladder wash — Participants will draw up the 45cc of normal saline into a 60cc syringe and instill via the intermittent catheter after the last catheterization prior to going to bed after trigger symptoms occur. Participants will be instructed to complete the USQNB-IC at the time of symptoms (in real time), and then continue completing the USQNB-IC at the determined frequency for the phase.
  Arms: Intravesical Bladder Wash (Prophylaxis Phase); Intravesical Bladder Wash (Treatment Phase)

SUMMARY:
This is the first ever comparative effectiveness study of an antibiotic-sparing novel self-management intervention to prevent complicated urinary tract infection (UTI).

DETAILED DESCRIPTION:
Urinary tract infection (UTI) is the most common outpatient infection world-wide, and for people with spinal cord injury (SCI) and neurogenic bladder (NB), it is the most common infection, secondary condition, cause for emergency room visits, and infectious cause of hospitalization. Despite its prevalence, attempts to ameliorate UTI among people with SCI are stymied by long-standing diagnostic challenges which arise from evidence gaps around "gold standard" diagnostic tests (urinalysis and urine culture) that have lower sensitivity and specificity for UTI in this population. A high prevalence of chronic inflammation leading to persistence of white blood cells (WBC) in the urine confounds the utility of WBC count, pyuria, and leukocyte esterase as biomarkers for UTI; nitrites in urine indicate the presence of only specific (but not all) organisms, many of which are present to a greater extent in the urine of people with SCI; and people with SCI have a high prevalence of asymptomatic bacteriuria. These physiologic changes render the gold standard diagnostic tests less useful for identifying UTI in persons with SCI.

SPECIFIC AIM 1 Compare the effects of Lactobacillus Rhamnosus GG (LGG®) + Saline bladder wash (BW) versus BW alone on USQNB-determined bladder (B1) and urine quality (B2) symptom burden (two co-primary outcomes) where participants self-manage in response to two trigger symptoms (cloudier and/or more foul-smelling urine).

SPECIFIC AIM 2 Compare the effects of LGG®+BW versus BW alone (in response to the two trigger symptoms) on key secondary outcomes: number of days lost from rehabilitation, work, and/or school; number of days symptomatic; number of interactions with the health care system due to urinary symptoms; exposure to antibiotics (days, volume).

SPECIFIC AIM 3 Compare the prophylactic effects of LGG®+BW versus BW alone on USQNB-determined bladder (B1) and urine quality (B2) symptom burden.

SPECIFIC AIM 4 Compare the prophylactic effects of LGG®+BW versus BW alone on key secondary outcomes: number of days lost from rehabilitation, work, and/or school; number of days symptomatic; number of interactions with the health care system due to urinary symptoms; exposure to antibiotics (days, volume).

SPECIFIC AIM 5 Compare satisfaction of participants who instilled LGG®+BW to satisfaction of those who instilled BW only and determine if dropouts are differentially attributable to either intervention being perceived by participants as "not working".

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. SCI at least 6 months duration;
3. NLUTD (as determined by their SCI physician or urologist);
4. Utilizing intermittent catheterization for bladder management; and
5. Community dwelling (discharged from the acute care setting).

Exclusion Criteria:

1. Known genitourinary pathology beyond neuropathic bladder (i.e., vesicoureteral reflux, bladder or kidney stones, etc.);
2. Use of prophylactic antibiotics;
3. Instillation of intravesical agents (e.g., gentamycin, saline; or Lactobacillus);
4. Immunodeficiency;
5. Any oral antibiotics within the past 2 weeks;
6. Psychologic or psychiatric conditions influencing the ability to follow instructions;
7. Participation in another study in which results would be confounded;
8. 6 months since prior exposure to intravesical LGG®; and
9. Active cancer (or within 5 years) or active autoimmune disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
International SCI Lower Urinary Tract Function Basic Data Set | Day 1
  A tool that describes urinary tract impairment, awareness of need to empty bladder, main bladder emptying method, medications used for bladder management, surgeries, and change in urinary symptoms in the past year. Score is not associated with outcome.
International SCI Core Data Set | Day 1
  Includes date of injury, dates of initial hospitalization admission and discharge, neurological data. Score is not associated with outcome.
NINDS Medical History CDE | Day 1
  A brief medical history using body system categories. Score is not associated with outcomes.
NINDS Prior and Concomitant Medications CDE | Day 1
  Contains whether or not the participant is taking a medication during the study protocol, name of the medication, reason for medication, medication dose, frequency, start and end dates, and free text. Score is not associated with outcomes.
Urinary Symptom Questionnaire for Neurogenic Bladder-Intermittent Catheter | (SA1 and SA3) Weekly up to 18 months
  Will measure change in urinary symptoms for those that use an intermittent catheter. Higher scores may mean worse outcomes.
Urinary Symptom Questionnaire for Neurogenic Bladder-Intermittent Catheter | (SA1) Day 1 post-instillation (Phase 2: treatment phase)
  Will measure change in urinary symptoms for those that use an intermittent catheter. Higher scores may mean worse outcomes.
Urinary Symptom Questionnaire for Neurogenic Bladder-Intermittent Catheter | (SA1) Day 2 post-instillation (Phase 2: treatment phase)
  Will measure change in urinary symptoms for those that use an intermittent catheter. Higher scores may mean worse outcomes.
Urinary Symptom Questionnaire for Neurogenic Bladder-Intermittent Catheter | (SA3) Twice weekly post-instillation for up to 6 months (Phase 3: prophylaxis phase)
  Will measure change in urinary symptoms for those that use an intermittent catheter. Higher scores may mean worse outcomes.
Patient Satisfaction Survey | At final USQNB-IC completion (between 13 to 18 months) or at participant drop-out
  We developed a simple three-item patient satisfaction "survey" that will be requested from only those individuals who used the intervention (LGG® +BW or BW only) at the time of final USQNB-IC completion, or at the drop out visit (for those who did use the intervention at least once). Participants will be asked to estimate, using a scale from 0% <totally dissatisfied/would absolutely never do this>, through 50% <neither satisfied nor dissatisfied/might do this> to 100% <completely satisfied/would absolutely always do this>:
  1. How satisfied with the intervention you used are you?
  2. Would you seek this intervention out and pay for it if insurance did not pay for it?
  3. Would you use or recommend the intervention in response to symptoms, prophylactically, or both? :At the drop out visit, we will ask these three questions and one additional item for those who used the intervention at least once, "Are you dropping out because the intervention was not working for you?"

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Groah, MD, MSPH, Principal Investigator — MedStar National Rehabilitation Hospital
Locations (1):
- MedStar National Rehabilitation Hospital, Washington D.C., District of Columbia, United States